CLINICAL TRIAL: NCT01926483
Title: A Prospective, Phase II Trial of a Trimodality Regimen for Stage III (N2) Non-small-cell Lung Cancer Using Concurrent Chemoradiotherapy as Induction Treatment Followed by Subsequent Resection
Brief Title: Phase II Trial of Regimen for Stage III (N2) NSCLC Using Induction Treatment Followed by Resection
Acronym: ZTOG-1202
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZTOG-1202
Record Dates: First submitted 2013-06-04; First posted 2013-08-21 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2012-07

CONDITIONS: Non-small Cell Lung Cancer Stage IIIA
Keywords: Stage IIIA-N2 NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Neoadjuvant Treatment (Experimental): Neoadjuvant Chemoradiotherapy
  Interventions: Other: Neoadjuvant Chemoradiotherapy

INTERVENTIONS:
Other: Neoadjuvant Chemoradiotherapy — Surgery followed by cisplatin-based regimen and concurrent radiation (46Gy/23f), consolidate the original regimen 2 cycles.

SUMMARY:
The investigators hypothesized that the Neoadjuvant Chemoradiotherapy was a beneficial treatment for Patients with Stage IIIA-N2 Non-Small Cell Lung Cancer, so we try to evaluate the security of treatment, the QoL of patients and the influence to the PFS and OS.

DETAILED DESCRIPTION:
Scheme:

Patients will receive different chemotherapy regimens depending on the pathological type.

Squamous cell carcinoma:Docetaxel/Cisplatin and concurrent radiation (46Gy/23f) followed by surgery, consolidate Docetaxel/Cisplatin 2 cycles.

Non-squamous cell carcinoma:Pemetrexed/Cisplatin and concurrent radiation (46Gy/23f) followed by surgery, consolidate Pemetrexed/Cisplatin 2 cycles.

ELIGIBILITY:
Inclusion Criteria:

* 18≤Age≤65;
* ECOG performance status of 0 or 1;
* Pathological diagnosis with Stage IIIA-N2 NSCLC which is clinically resectable and the N2 is diagnosed by either mediastinoscopy,EBUS,PET/CT;
* WBC≥4.0×109/l, ANC≥1.5×109/l, PLT≥100.0×109/l, Hb≥90g/l;hepatorenal function is normal;
* Without a history of other malignancies before enrollment, except for non-melanoma skin cancer, in situ cervical cancer;
* The patient can understand the research and sign the informed consent.

Exclusion Criteria:

* Female in pregnancy or lactating;Female of childbearing age without contraception;
* With acute infection or other serious underlying disease;
* With a significant history of neurological of psychiatric disease，including the dementia which may affect the ability to understand and sign the informed consent;
* Have received other treatment within the last 30 days before enrollment;
* With uncontrollable diabetes(blood glucose is unstable after treatment or FBG≥8mol/L).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
PFS | up to 3 years

SECONDARY OUTCOMES:
Adverse events | participants will be followed for the duration of hospital stay,an expected average of 100 days and every 3 months thereafter for 5 years
  observe and record the toxicity profile(including but not limit to mucositis,liver and kidney function,et al.)according NCI-CTCAE(3rd edition) during the neoadjuvant chemoradiation and follow-up.
QOL | up to 3 years
OS | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Weimin Mao, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China